CLINICAL TRIAL: NCT05365880
Title: Sphenopalatine Ganglion Block for the Treatment of Post-Stroke Headache
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to COVID-19 and both co-investigators have departed from the institution, we weren't able to enroll participants. Additionally, funding has lapse
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 138103
Record Dates: First submitted 2022-04-25; First posted 2022-05-09 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Headache; Stroke; Ischemic Stroke
Keywords: Post-Stroke Headache; Sphenopalatine Ganglion (SPG) block
MeSH Terms: conditions — Headache; Stroke; Ischemic Stroke; Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liquid Lidocaine (Experimental): The investigational treatment is 1.5 mL of aqueous 2% lidocaine.
  Interventions: Drug: Liquid Lidocaine
- Sham Placebo (Placebo Comparator): The placebo arm is 1.5mL of aqueous of saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liquid Lidocaine — The investigational treatment is 2 mL of aqueous 2% lidocaine.
  Arms: Liquid Lidocaine
Drug: Placebo — The active placebo comparator will be provided to participant.
  Arms: Sham Placebo

SUMMARY:
Determine the effects of sphenopalatine ganglion (SPG) block in post-stroke headache.

DETAILED DESCRIPTION:
The purpose of this study is to determine if sphenopalatine ganglion (SPG) block is a safe and effective treatment for acute post-stroke headache. Current literature lacks randomized controlled studies regarding the efficacy of different treatment modalities for acute post-stroke headache; additionally, there are no evidence-based guidelines for the treatment of acute post-stroke headache. Sphenopalatine ganglion block is a non-invasive procedure where an anesthetic agent is injected into the nares, reaching the SPG to relieve pain and autonomic features. This treatment has been effective in a variety of headache types but to our knowledge has not been studied in acute post-stroke headache.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older;
2. hospitalization at the University of Utah Hospital with a diagnosis of acute ischemic or hemorrhagic stroke; confirmed acute post-stroke headache by treating physician;
3. meets at least one of the following International Classification of Headache Disorder-3 (ICHD-3) criteria: 6.1.1.1 (Acute Headache Attributed to Ischemic Stroke), 6.2.1 (Headache attributed to non-traumatic intracerebral hemorrhage), 6.2.2 (Acute headache attributed to non-traumatic subarachnoid hemorrhage); received at least one medication for headache during hospitalization.

Exclusion Criteria:

1. Previous treatment with SPG Block for post-stroke headache
2. history of prophylactic medication use for headache or migraine;
3. pregnant at time of stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-03-22 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Migraine Headaches During Treatment Phase | 90 days
  Evaluate the efficacy of Lidocaine delivered to SPG, based on the use of rescue medication and number of headache in headache diary

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 90 days
  The quantitative scale ranges from 0 to 10, with 0 meaning "no headache at all" and 10 meaning "the worst possible headache."
Adverse effect | 90 days
  Bitter taste, nose bleeding, throat discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Adam H de Havenon, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delpont B, Blanc C, Osseby GV, Hervieu-Begue M, Giroud M, Bejot Y. Pain after stroke: A review. Rev Neurol (Paris). 2018 Dec;174(10):671-674. doi: 10.1016/j.neurol.2017.11.011. Epub 2018 Jul 24. PMID 30054011
- [Result] Lai J, Harrison RA, Plecash A, Field TS. A Narrative Review of Persistent Post-Stroke Headache - A New Entry in the International Classification of Headache Disorders, 3rd Edition. Headache. 2018 Oct;58(9):1442-1453. doi: 10.1111/head.13382. Epub 2018 Aug 27. PMID 30152015
- [Result] Ho KWD, Przkora R, Kumar S. Sphenopalatine ganglion: block, radiofrequency ablation and neurostimulation - a systematic review. J Headache Pain. 2017 Dec 28;18(1):118. doi: 10.1186/s10194-017-0826-y. PMID 29285576
- [Result] Rosso C, Felisati G, Bulfamante A, Pipolo C. Cluster headache: crosspoint between otologists and neurologists-treatment of the sphenopalatine ganglion and systematic review. Neurol Sci. 2019 May;40(Suppl 1):137-146. doi: 10.1007/s10072-019-03796-5. PMID 30877613
- [Result] Androulakis XM, Krebs KA, Ashkenazi A. Hemicrania continua may respond to repetitive sphenopalatine ganglion block: A case report. Headache. 2016 Mar;56(3):573-9. doi: 10.1111/head.12783. Epub 2016 Mar 1. PMID 26926875
- [Result] Harriott AM, Karakaya F, Ayata C. Headache after ischemic stroke: A systematic review and meta-analysis. Neurology. 2020 Jan 7;94(1):e75-e86. doi: 10.1212/WNL.0000000000008591. Epub 2019 Nov 6. PMID 31694924
- [Result] Mulder IA, Li M, de Vries T, Qin T, Yanagisawa T, Sugimoto K, van den Bogaerdt A, Danser AHJ, Wermer MJH, van den Maagdenberg AMJM, MaassenVanDenBrink A, Ferrari MD, Ayata C. Anti-migraine Calcitonin Gene-Related Peptide Receptor Antagonists Worsen Cerebral Ischemic Outcome in Mice. Ann Neurol. 2020 Oct;88(4):771-784. doi: 10.1002/ana.25831. Epub 2020 Aug 7. PMID 32583883
- [Result] Levin M. Opioids in headache. Headache. 2014 Jan;54(1):12-21. doi: 10.1111/head.12266. PMID 24127913
- [Result] Cady R, Saper J, Dexter K, Manley HR. A double-blind, placebo-controlled study of repetitive transnasal sphenopalatine ganglion blockade with tx360((R)) as acute treatment for chronic migraine. Headache. 2015 Jan;55(1):101-16. doi: 10.1111/head.12458. Epub 2014 Oct 23. PMID 25338927
- [Result] Maizels M, Scott B, Cohen W, Chen W. Intranasal lidocaine for treatment of migraine: a randomized, double-blind, controlled trial. JAMA. 1996 Jul 24-31;276(4):319-21. PMID 8656545